CLINICAL TRIAL: NCT04927520
Title: Safety and Efficacy of Treatment for Middle Cerebral Artery Aneurysms: a Prospective and Multicenter Trial
Brief Title: Prospective, Multicenter Cohort Study on the Safety and Efficacy of Treatment for Middle Cerebral Artery Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Jinhua Central Hospital (Other); Ningbo No. 1 Hospital (Other); The Central Hospital of Lishui City (Other); Taizhou Hospital (Other); People's Hospital of Quzhou (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-174
Record Dates: First submitted 2021-06-05; First posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Middle Cerebral Artery Aneurysm
Keywords: Middle cerebral artery aneurysms; Clipping surgery; Coil embolization; Endovascular therapy; Unruptured aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular therapy group: Unruptured middle cerebral artery aneurysms treated with coil embolization
- Clipping surgery group: Unruptured middle cerebral artery aneurysms treated with clipping surgery

SUMMARY:
Intracranial aneurysm is one of the most common cerebrovascular diseases, with a prevalence of about 3.2%. With the aging of the population and the further popularization of MRA and other examination methods, the prevalence of intracranial aneurysm will further increase. Rupture of intracranial aneurysm is an important cause of death and severe disability in patients. The annual rate of rupture of intracranial aneurysm is about 1%, and the size of aneurysm, the location of aneurysm in the posterior circulation, and the history of subarachnoid hemorrhage on the aneurysm wall are the risk factors for aneurysm rupture. Phases are currently recognized tools for assessing the risk of aneurysm rupture, which can provide important guidance for neurosurgeons and patients to decide whether to actively intervene. In the last century, for patients with intracranial aneurysm with high risk of rupture, craniotomy and clipping for intracranial aneurysm was the gold standard for treatment.

However, with the rapid development of embolization technology and materials in the past 20 years, the application of endovascular embolization for intracranial aneurysms has been more and more widely, especially after several large prospective studies such as ISAT and ISUIA, endovascular embolization has more advantages over craniotomy clipping.Whereas, it is still very popular to adopt craniotomy clipping for middle cerebral artery aneurysms, the main reasons for which are relative superficial location, wider aneurysm neck, smaller parent artery and more branching vessels, etc., which make early endovascular embolization treatment not advantageous. With the maturity of stent-assisted embolization technology in recent years, the use of a new generation of stents, and the improvement of perioperative anti-platelet strategies, endovascular embolization has achieved good results in the treatment of middle artery aneurysms. However, these studies were retrospective, single-center studies, subject to a variety of confounding factors, and the reliability of the results is limited.

Therefore, it will be of great clinical significance to carry out a prospective, multi-center clinical study on the treatment strategy of middle cerebral artery aneurysms.

Patients with unruptured middle cerebral artery aneurysms who had been diagnosed with at least one imaging （CTA/MRA/DSA）were enrolled. The treatment including endovascular embolization and craniotomy clipping was determined according to routine management in the center. After receiving informed consent from the patients, the safety and effectiveness data were obtained to verify whether endovascular embolization was safe and effective. Through further follow-up and data analysis, protective factors and risk factors for the treatment of middle cerebral artery aneurysms were investigated. Through well-designed clinical studies, safer and more effective treatment methods can be found, and potential factors leading to perioperative complications can be found, ultimately improving the prognosis of patients with middle cerebral artery aneurysms.

DETAILED DESCRIPTION:
1. Data collection and management A unified and open public health platform will be established, and data will be centrally recorded in each central unit for verification by inspectors. An open network data platform for intracranial aneurysm research was established by the management personnel of different qualification levels. In order to ensure the advancement and sustainable development of the data platform construction, a public research platform for intracranial aneurysms shared in the province was built by using the keywords and retrieval items commonly used in China.

   After researcher training and standardized study of the scheme, the formal trial was started. A team of experts will be selected to form an inspection team, which will initiate visits to each organization and conduct the first inspection visit as soon as possible after screening the first subject. Regular monitoring visits are required until the end of the experiment. All the data were collected according to the electronic medical record (CRF) form, and then the aneurysm data (EDC) was managed according to the CRF form, and the accuracy and rigor of the data were checked in time.

   This study establishes a management committee, including clinical experts, evidence-based medicine experts, and CRO clinical study supervisors, who are responsible for project design, task formulation, supervision of project implementation, data analysis and formulation of standards and guidelines.

   The central laboratory and imaging interpretation center were established to carry out unified standard central storage for clinical specimens. The unified image and laboratory technology platform can be used for the image examination and post-processing technology in the project. Uniform standard interpretation of imaging data was carried out. A unified, standardized and efficient transmission mechanism for clinical specimens, data and data in each center was established.

   Establish a data management committee, set up a network data platform and be responsible for the construction and maintenance of the database, conduct real-time supervision on the quality of the input data, ensure the safety, integrity and accuracy of the data, establish and organize the implementation of the platform or offline dual-channel error correction and reminder mechanism. Set and manage the rights of all project participants on the data platform, monitor and record the data entry, modification and retrieval, set and manage the data publication of the open platform. Contact and consult statistical experts to conduct periodic analysis of data results and generate research reports.

   Relying on professional CRO company, in the implementation process for the implementation of the progress and quality of the implementation of random inspection supervision. At the same time, set up a data regular self-check mechanism. Establish a mechanism for regular training and evaluation of research participants. During the research progress, regular project coordination meetings were held to timely coordinate and solve problems in the process of the project.
2. Sample size Sample size was calculated according to a calculation formula (α=0.05, bilateral test, 80% assurance). According to the literature and the data of the center, the rate of MRS<2 at 3 months was 95% for patients with endovascular interventional, and was 85% for those with craniotomy and clipping. The number of samples needed for each group was calculated by the software PASS15 to be at least 141. Considering that the maximum shedding rate of 20% might occur during the clinical follow-up, 180 cases were needed for each group, and 360 subjects were finally decided to be included in the study.
3. Statistical Methods Statistical analysis of planned primary and secondary study endpoints will be conducted in accordance with the intentionality treatment principle. Subgroup analysis According to the needs of the experiment, the subjects can be divided into different centers, male and female, and different age groups for corresponding subgroup analysis. Methods for processing lost data Statistical analysis did not follow the study protocol population definition and other statistical methods were used to deal with lost data (e.g. multiple interpolation).
4. Ethical approval of clinical research projects The study plan was reviewed and approved by the Ethics Committee of the Second Affiliated Hospital of Zhejiang University School of Medicine. The study protocol was designed and implemented in accordance with the International Conference on Harmonization for Good Clinical Practice (ICH-GCP) guidelines. In line with the national ethical behavior requirements, applicable to local laws and regulations, in strict compliance with the World Medical Association (WMA) Declaration of Helsinki ethical provisions.
5. Informed Consent Process Improve the relevant examinations, check the inclusion and exclusion criteria of patients, and send the detailed information of the study to patients or their legal clients. If the patients or legal clients agree to participate in the study, they need to sign two copies of informed consent. The original consent form should be kept in the patient's study folder and another copy given to the patient. Patients or legal clients have the right to terminate their participation in the study at any time, and their decision will be recorded in the patient's study record.
6. confidentiality The investigators will take every step to respect the privacy of the participants in the study. Only data that does not contain identifying information will be entered into the central research database to ensure the privacy of participants. In the process of monitoring data quality and study protocol compliance, the data monitor will refer to the medical records of the subject's clinical center and record them on the patient information sheet. In the reporting data and results, all personal information and research center information will be hidden to protect the privacy of participants.
7. Adverse events management Adverse events occurred in the process of adverse events refers to the study of the subjects has a harmful effect on the health of all events. Serious Adverse Event Category: Serious Adverse Event refers to any event that occurred during the course of the study that had a serious adverse effect on the health of the subjects. Include: cause the subject to be hospitalized, prolong the length of the subject's hospital stay, cause the subject to be disabled, cause the subject's neurological or physical dysfunction, cause the subject's offspring to be born with a deformity, endanger the subject's life, the subject's death or other events that have a serious adverse effect on the subject's health. Adverse events reported to process all kinds of adverse events: take timely measures to deal with, and recorded in a report on the case. Serious adverse event (SAE) : take timely measures to deal with, and recorded in a report on the case, the researchers decided to withdrawal or by drugs, immediately report ethics committee, the drug clinical trial institution and the sponsor, 24 hours, report to the national and provincial food and drug administration. SAE is required to report adverse events and proximate errors via the Intra-hospital Network Notification System.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 middle cerebral artery aneurysm confirmed by imaging (CTA/MRA/DSA);
* Accept endovascular intervention or middle cerebral artery aneurysm clip craniotomy, regardless of whether there is a clinical symptoms;
* Multiple aneurysms, whether usual treatment, but it requires the treatment time interval to > 6 months;
* The subjects currently has independent life ability, namely the mRS score 3 points or less;
* The patient or family agreed to sign a consent form.

Exclusion Criteria:

* Patients with other intracranial vascular malformations, such as AVM and AVF;
* Fusiform, traumatic, bacterial or dissecting aneurysm;
* Ruptured middle cerebral artery aneurysm associated with intracranial hematoma;
* Intracranial or other parts of the patients with malignant tumors;
* General condition is bad, is expected to survival time less than 1 year or poor body condition, can't tolerate anesthesia or aneurysm surgery patients;
* Involved with other intracranial aneurysm patients clinical research;
* A hospital surgery clip or endovascular treatment of patients at the same time;
* Refused to follow-up of patients.

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed unruptured middle artery aneurysm and treated with coil embolization or endovascular therapy
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-06-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
mRS at 3 months | at 3 months
  the favorable outcome was defined as mRS 0-2
Complication | during hospitalization up to 14 days
  including aneurysm rupture, aneurysm recurrence, stroke and other cerebrovascular disease

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China